CLINICAL TRIAL: NCT04903223
Title: Effects of Pediatric Liver Adiposity on Statin Disposition and Response
Brief Title: Liver Adiposity Effects on Pediatric Statin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Jon Wagner, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001550
Record Dates: First submitted 2021-05-17; First posted 2021-05-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cholesterol; Lipidosis
MeSH Terms: conditions — Lipidoses | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label, prospective, investigation to quantify the effects hepatocellular fat has on hepatic statin transport (SA1) and response (SA2) in children and adolescents.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Baseline Mevalonate and MRI Imaging (No Intervention)
- Mevalonate Change After Rosuvastatin (Experimental)
  Interventions: Drug: Rosuvastatin 10mg

INTERVENTIONS:
Drug: Rosuvastatin 10mg — Rosuvastatin will be administered to all participants on Study Day #2
  Arms: Mevalonate Change After Rosuvastatin

SUMMARY:
Single center, open-label, prospective investigation to quantify the effects hepatocellular fat has on hepatic statin transport and response in children and adolescents in obese and non-obese children and adolescents 8-21 years of age with normal, wild-type SLCO1B1 c.521TT genotype that are dosed rosuvastatin

ELIGIBILITY:
Inclusion Criteria:

* 8-21 years
* LDL cholesterol >130mg/dl (>95% percentile)
* SLCO1B1 c.521TT genotype
* Provide informed permission-assent(<18 yrs.) or consent (≥18 yrs.)
* Fasting overnight (~8 hrs.)
* Enrolled in Cardiology Pharmacogenomic Repository

Exclusion Criteria:

* Pregnancy
* Non-fasting
* Non-removable metal in body or MRI unsafe
* Currently on statin therapy and unwilling to wash out of statin therapy for at least 4 weeks prior to Visit 1 and throughout the duration of the study.
* Underlying unrepaired congenital or acquired cardiovascular defects or repaired congenital or acquired cardiovascular defects with hemodynamically significant residual disease.
* History of underlying or laboratory evidence of underlying intestinal, metabolic, autoimmune, renal disease that can alter rosuvastatin disposition* (absorption, metabolism, distribution, or clearance)
* Pharmacotherapy that interacts with statins (OATP1B1 inducers/inhibitors) *
* Inability to swallow a tablet
* >5x the age-specific upper limit of normal for AST, ALT, total and conjugated bilirubin
* Diarrhea in the last 24 hours
* Anything that would exclude a participant from completing an MRI, such as pacemakers, claustrophobia, or body habitus (e.g., weight greater than 350 lbs.)

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate effect of Liver Fat Percentage (on MRI) on AUC | 2 years
  We expect that increased liver adiposity will be associated with higher systemic statin exposure and thus, place those with higher liver adiposity fraction at increased risk for drug toxicity.
Evaluate effect of Liver Fat Percentage (on MRI) on change on plasma mevalonate level | 2 years
  We expect that increased liver adiposity will be associated with an attenuated mevalonate response to a statin in obese children placing those with increased liver adiposity at risk for treatment failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States